CLINICAL TRIAL: NCT00188370
Title: Ultrasound Biomicroscopy for Monitoring Apoptosis in Lymphoma, Melanoma and Basal Cell Carcinoma Patients During Chemotherapy or Radiation Therapy
Brief Title: Ultrasound Biomicroscopy - Apoptosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UHN REB 01-0508-C
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-09

CONDITIONS: Lymphoma; Lymphoma, Non-Hodgkin; Melanoma; Carcinoma, Basal Cell
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Melanoma; Carcinoma, Basal Cell

INTERVENTIONS:
Procedure: high frequency ultrasound imaging

SUMMARY:
A group of researchers at the Ontario Cancer Institute/Princess Margaret Hospital have discovered that a very specific form of cell death 'apoptosis' can be detected using high-frequency ultrasound imaging. This type of cell death is recognized to occur in tumours in response to various different chemotherapeutic drugs and in response to radiation therapy. This group of researchers has confirmed that high-frequency ultrasound can detect apoptosis in response to tumour treatments experimentally using cell culture and experimental animal systems. The ultrasound approach is now being evaluated clinically in a 3-year clinical trial enrolling a target of 200 patients including Hodgkin's disease and non-Hodgkin's disease lymphoma patients, melanoma patients and patients with basal cell carcinoma. Our hope is to be able to use this type of imaging system in the future to clinically monitor the effects of therapy on tumours and rapidly detect tumours which are not responding so that changes in therapy can be made much quicker than presently possible.

ELIGIBILITY:
Inclusion Criteria:

* lymphoma patients with superficial lesions prior to starting chemotherapy or after relapse of disease
* patients with superficial melanoma lesions
* patients with superficial basal cell carcinoma lesions
* Informed consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 1999-04; Study Completion 2004-12

PRIMARY OUTCOMES:
Feasibility study of the use of Ultrasound Biomicroscopy for monitoring tumour response of lymphoma and melanoma patients to chemotheapy or radiation therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Tsang, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada